CLINICAL TRIAL: NCT05366803
Title: Women's Health Initiative Strong and Healthy Silent Atrial Fibrillation Recording Study
Brief Title: Women's Health Initiative Silent Atrial Fibrillation Recording Study
Acronym: WHISH STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marco Perez, Associate Professor of Medicine (Cardiovascular Medicine), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 40082
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Intervention (Experimental): The Physical Activity Intervention Group will receive guidance on being physically active, including aerobics, flexibility, balance, strength, and decreased sedentary time. The primary resource is the National Institute of Aging Go4Life exercise and physical activity materials. The materials are based on the United States national guidelines for physical activity for older adults. Participants will wear the Zio patch monitor (electrocardiographic loop monitoring device) for 8 days at baseline, as well as at 6 months and again at one year, for a total of 3 times.
  Interventions: Behavioral: Physical Activity
- Usual Activity Control (No Intervention): Participants will wear the Zio patch monitor (electrocardiographic loop monitoring device) for 8 days at baseline, as well as at 6 months and again at one year, for a total of 3 times. Participants carry about their normal activities during this period.

INTERVENTIONS:
Behavioral: Physical Activity — The PA intervention will consist of a multimodal activity program of aerobics, balance, strength, flexibility. The intervention will involve encouraging participants to increase all forms of PA throughout the day and to decrease sedentary time, such as sitting. This may include activities such as leisure sports, gardening, use of stairs instead of escalators, leisurely walks with friends, and less use of remote control devices.The intervention is conducted primarily by mail with website support and resources available.
  Arms: Physical Activity Intervention

SUMMARY:
The purpose of the WHISH STAR study is to investigate whether or not those who are randomized to exercise intervention have higher rates of atrial fibrillation on review of medical records and, in a subset, on screening with a cardiac ECG patch monitor. We will also study whether those with a known history of AF have any changes in AF hospitalizations due to exercise.

DETAILED DESCRIPTION:
The Silent Atrial Fibrillation Recording study (STAR) study is an ancillary study of the NIH-funded Women's Health Initiative Strong and Healthy (WHISH). The purpose of the Women's Health Initiative Strong and Healthy study (WHISH) is to investigate if light to moderate exercise decreases incident atrial fibrillation (AF) among women over 65 who have no baseline AF. The purpose of the STAR study is to investigate the effect of exercise intervention on incident atrial fibrillation ascertained with diagnostic codes. In a subset of women, subclinical atrial fibrillation will be ascertained with cardiac patch ECG monitoring technology (iRhythm's ZIO® XT Patch). This subgroup of WHISH study participants will undergo an 8 day cardiac patch recording at baseline, six (6) months, and one (1) year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects already enrolled in the parent WHISH study.
* Subjects who are at high risk of developing atrial fibrillation.

Exclusion Criteria:

* Subjects who have had atrial fibrillation at baseline.

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — The participants are all older women, since the parent study is a post-menopausal study from the Women's Health Initiative.
Enrollment: 1257 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Incidence of Atrial Fibrillation Due to Exercise | One year
Number of Participants without Clinically Diagnosed Atrial Fibrillation (AF) Found to have Silent AF with Prolonged ECG Patch Monitoring | One year

CONTACTS AND LOCATIONS:
Overall Officials: Marco Perez, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Lin JY, Larson J, Schoenberg J, Sepulveda A, Tinker L, Wheeler M, Albert C, Manson JE, Wells G, Martin LW, Froelicher V, LaMonte M, Kooperberg C, Hlatky MA, Greenland P, Stefanick ML, Perez MV. Serial 7-Day Electrocardiogram Patch Screening for AF in High-Risk Older Women by the CHARGE-AF Score. JACC Clin Electrophysiol. 2022 Dec;8(12):1523-1534. doi: 10.1016/j.jacep.2022.08.024. Epub 2022 Oct 26. PMID 36543503